CLINICAL TRIAL: NCT04659005
Title: Pilot Testing and Evaluation of a Nurse-led Decision Counseling Program to Improve Decision-making and Uptake of Hepatocellular Carcinoma Screening Among Patients With Hepatitis B Virus Infection: A Randomized Controlled Trial
Brief Title: Nurse-led Decision Counseling on Hepatocellular Carcinoma Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, LI Caixia, Ms., Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: cuhknurs01
Record Dates: First submitted 2020-10-31; First posted 2020-12-09 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B; Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepatitis B; Screening; Early detection; Nurse-led intervention; Decision counseling
MeSH Terms: conditions — Hepatitis B; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-led decision counseling group (Experimental): Provide education, tailored information, decision support, and psychosocial support regarding hepatocellular carcinoma screening
  Interventions: Other: Nurse-led decision counseling
- Control group (Other): Usual care provided by the hospital, including one-page written education information about diet, medications, and daily exercises.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Nurse-led decision counseling — Provide education, tailored information, decision support, and psychosocial support regarding hepatocellular carcinoma screening
  Arms: Nurse-led decision counseling group
Other: Usual care — Usual care provided by the hospital, including one-page written education information about diet, medications, and daily exercises
  Arms: Control group

SUMMARY:
Hepatocellular carcinoma (HCC) is a common malignancy with poor prognosis worldwide. The asymptomatic of early-stage HCC may lead most patients diagnosed at advanced stages. This highlights the importance of HCC screening among high-risk populations to detect HCC at early stages and achieve better survival. Hepatitis B virus (HBV) infection is a major cause of HCC in China, but the utilization of HCC screening is suboptimal among patients with HBV infection.

Currently, there are no-theory based intervention, to our knowledge, has been reported to improve HCC screening decision-making and uptake among patients with HBV infection . Therefore, based on our previous systematic review, the current study has proposed a nurse-led decision counseling program to improve decision-making and uptake of HCC screening among patients with HBV infection in mainland China.

Participants in intervention group will receive nurse-led decision counseling. The intervention components include 40-minute education and tailored information regarding HCC screening. At the second week, decision support will be provided through 30-minute telephone call. At the third week, another telephone call (20 minutes) will be provided to help participants identify and address barriers to HCC screening.

Participants in control group will receive usual care. After the intervention and at 3-month follow-up, the study will collect data related to HCC screening uptake rates. Findings are paramount to promote informed choice in HCC screening and early HCC detection to improve survival outcomes among patients with HBV infection.

DETAILED DESCRIPTION:
Participants in the intervention group will receive the following three-week, three-session intervention. The details are as follows.

Education (20 min). At first week, education will be delivered through face-to-face for the following information: (1) HBV infection and increased HCC risk; (2) HCC screening recommendations regarding eligibility, available screening tests and recommended screening intervals; (3) pros/advantages of undergoing HCC screening; (4) cons/disadvantages or uncertainties of undergoing HCC screening; (5) implications of positive screening results; and (6) health costs. The education material will be present in a self-made manual, which will be explained and distributed to each participant.

Tailored psychosocial information (20 min). It will be conducted after education. The tailored messages will be developed to form a message library for each sub-scale of the preventive health model instrument with scoring ≤ 3 and > 3. The contents will be based on HCC screening guidelines and recommendations. The nurse counsellor will select and explain tailored information based on individual's responses to the preventive health model instrument.

Values clarification exercises (30 min). At the second week, the decision counselor will work with participants through telephone-based way to go through values clarification exercises, in which participants will: (1) review the listed pros and cons decision factors of undergoing HCC screening one by one; (2) indicate the extent to which each pros and cons matters to them by giving stars; (3) add any other reasons for choosing or not choosing HCC screening and indicate their importance; and (4) indicate their decision preferences toward undergoing HCC screening, unsure, or not undergoing HCC screening.

Exploring and addressing implementation barriers (20 min). At the third week, the decision counselor will work with participants, through telephone-based ways, to explore possible barriers to undertake HCC screening; identify possible solutions or available resources to the identified barriers via brainstorming; and encourage implementation of the chosen solution to overcome the barriers and schedule for HCC screening.

ELIGIBILITY:
Inclusion Criteria:

* patients with HBV infection (HBsAg positive), aged 18-65 years old
* have been recommended to have HCC screening, including liver cirrhosis, males over age 40, women over age 50, and family history of HCC
* can understand Chinese
* without an liver ultrasound or serum alpha-fetoprotein test in the previous six months at the time of inclusion

Exclusion Criteria:

* have comorbid condition, including co-infection with hepatitis C, human immunodeficiency virus, and alcoholic liver disease
* have hepatocellular carcinoma diagnosis
* have undergone liver transplantation
* have encephalopathy
* not willing to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
HCC screening uptake rates | Immediately after intervention and three months after intervention
  The liver ultrasound, serum alpha-fetoprotein, dynamic computed tomography, and magnetic resonance are all considered as screening tests in the current study.

SECONDARY OUTCOMES:
HCC screening knowledge questionnaire | Baseline, immediately after intervention and three months after intervention
  It will be developed to measure knowledge regarding HCC and HCC screening recommendations. The yes or no questions and multiple-choice questions will be used to rate participants' responses by giving one point for a correct answer and zero point for an incorrect answer.
Preventive health model construct instrument. | Baseline, immediately after intervention and three months after intervention
  It has five domains with 16 items measuring salience and coherence (four items), cancer worriers (two items), perceived susceptibility (four items), response efficacy (two items), and social influence (four items).
Decisional conflict scale | Baseline, immediately after intervention and three months after intervention
  It consists of five subscales, including uncertainty, feeling informed, clarify related to personal values, feeling supported, and effective decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: Caixia Li, Principal Investigator — The Nethersole School of Nursing, The Chinese University of Hong Kong
Locations (2):
- China (2):
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The Nethersole School of Nursing, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li C, Lu X, Xu J, Gao F, Lee E, Chan CWH. Effectiveness of a nurse-led decision counselling programme on hepatocellular carcinoma screening uptake among patients with hepatitis B: A randomised controlled trial. Int J Nurs Stud. 2023 Dec;148:104610. doi: 10.1016/j.ijnurstu.2023.104610. Epub 2023 Sep 21. PMID 37801936
- [Derived] Li C, Lu X, Gao F, Lee E, Chan CWH. Development of a nurse-led decision counseling program for improving hepatocellular carcinoma screening: A typology-guided feasibility study. Asia Pac J Oncol Nurs. 2023 Mar 9;10(6):100215. doi: 10.1016/j.apjon.2023.100215. eCollection 2023 Jun. PMID 37305610
- See also: Our published review used to develop the current intervention and titled: Effects of nurse-led interventions on early detection of cancer: A systematic review and meta-analysis — https://doi.org/https://doi.org/10.1016/j.ijnurstu.2020.103684